CLINICAL TRIAL: NCT03117075
Title: The Efficacy of Pain Management With Self-reporting Pain Monitoring
Brief Title: The Efficacy of Pain Management With Self-reporting Pain Monitoring System in Cancer Patient
Acronym: pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: DERSHENG SUN (Other)
Responsible Party: Sponsor-Investigator, DERSHENG SUN, clinical assistant professor, The Catholic University of Korea
Organization: The Catholic University of Korea (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: XC15EIMI0099KUD
Record Dates: First submitted 2016-01-19; First posted 2017-04-17 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Pain
Keywords: cancer pain, wearable device
MeSH Terms: conditions — Pain; Cancer Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): using device for scoring pain scale, named "ANAPA®"
  Interventions: Device: using device for scoring pain scale, named "ANAPA®"

INTERVENTIONS:
Device: using device for scoring pain scale, named "ANAPA®" — wearable device for scoring pain scale

SUMMARY:
To compare the pain scales between clinician evaluated and reported with wearable device by patients.

DETAILED DESCRIPTION:
To compare the pain scales between clinician evaluated and reported with wearable device by patients with cancer of advanced stage.

ELIGIBILITY:
Inclusion Criteria:

* over 20 year old
* cancer pain with visual analog scale or numeric rating scale score >/- 4
* opioids candidates
* with informed consent form

Exclusion Criteria:

* life expectancy within 3 months

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2017-05-15 (Estimated); Primary Completion 2017-11-14 (Estimated); Study Completion 2018-04-14 (Estimated)

PRIMARY OUTCOMES:
Actual difference of pain scales | 1 week after using wearable pain scale device - baseline and 1 week.
  comparing the pain scale assessed by wearable device and that assessed by physician when out patient clinic.

CONTACTS AND LOCATIONS:
Overall Officials: YOONHO KO, MD, PhD, Principal Investigator — Uijeongbu St. Mary's Hospital, The Catholic University of Korea
Locations (2):
- South Korea (2):
  - Daejeon St. Mary's Hospital, the Catholic University of Korea, Daejeon
  - Seoul St. Mary's Hospital, the Catholic University of Korea, Seoul

IPD SHARING:
Plan to Share IPD: No